CLINICAL TRIAL: NCT00804739
Title: Adapting Collaborative Care Perinatal Depression Treatment to a Pediatric Setting - Pilot Phase
Brief Title: Perinatal Depression Treatment in a Pediatric Setting- Pilot Phase
Acronym: MITT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Linda Chaudron, Associate Professor, Department of Psychiatry, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R34MH082141-01 (NIH)
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Postpartum Depression
Keywords: Major Depression; Postpartum Depression; Perinatal Depression; Treatment Feasibility; Treatment Engagement; Treatment Adherence; Postpartum; Interpersonal Psychotherapy; IPT; Sertraline; Zoloft
MeSH Terms: conditions — Depression, Postpartum; Depressive Disorder, Major; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MITT (Experimental): Mothers will be assigned to the Mother-Infant Treatment Team (MITT)and will receive either psychotherapy or sertraline or both as well as outreach.
  Interventions: Other: Mother-Infant Treatment Team

INTERVENTIONS:
Other: Mother-Infant Treatment Team — This is a treatment team approach that allows for outreach. The clinical team will be a nurse practitioner of psychiatry and a social worker. The nurse practitioner will provide either interpersonal psychotherapy, sertraline or both as indicated.

SUMMARY:
The purpose of this project is to test whether a new model of collaborative care depression treatment adapted to the needs and preferences of low-income, urban mothers with perinatal depression and to a pediatric clinic setting increases engagement in and adherence to perinatal depression treatment.

DETAILED DESCRIPTION:
This research project consists of two phases that are designed, in sequence, to adapt standard collaborative care depression treatment to the unique needs of low-income depressed postpartum women and to the pediatric setting where women will receive the treatment. These adaptations, in turn, are designed to improve maternal engagement in and adherence to depression treatment, the primary outcomes at this early stage of intervention development. Phase I is the initial pilot project in which the model will be developed. We will 1) adapt standard collaborative care depression models into the Mother-Infant Treatment Team (MITT) intervention and develop a procedure manual based on maternal and provider input, 2) pilot the MITT intervention with 10 depressed mothers to test the feasibility of implementing the model, and 3) evaluate the experiences of participating mothers and providers to revise and finalize MITT processes and procedures.

Phase II will be an open label trial of MITT to determine whether MITT is associated with improved maternal engagement and adherence to depression treatment.

We will pilot MITT with 10 mothers to determine the feasibility of implementing MITT. We will collect recruitment and logistical feasibility measures. We will also determine engagement and adherence rates to treatment as well as the effort required to engage women in treatment.

We will determine mothers' and providers' perceptions of their experiences with MITT and will use all of this information to revise the MITT protocol in preparation for Phase II.

ELIGIBILITY:
Inclusion Criteria:

1. Mothers of infants 12 months of age or younger who present to the Pediatric Practice at Golisano Children's Hospital
2. Women who are 18 years of age or older
3. Mothers who understand and speak English sufficiently to participate in therapy with an English speaking provider
4. Have a current score of > 10 on the EPDS
5. Provide written informed consent
6. Meet criteria for unipolar major depressive disorder.

Exclusion Criteria:

Women who:

1. do not speak or understand English well enough to participate in the therapy with an English speaking provider
2. are under 18 years of age
3. children are not cared for at the Pediatric Practice at the Golisano Children's Hospital
4. are actively psychotic, suicidal or homicidal,
5. require treatment (including additional psychotropic medications) not provided by MITT,
6. in the judgment of the MITT psychiatric provider require a higher level of psychiatric care (i.e. partial hospitalization, hospitalization, intensive case management),
7. are in active counseling or psychotherapy,
8. are under the care of a psychiatric provider and/or are receiving active treatment for depression including light therapy, ECT, or antidepressants
9. are receiving psychotropic medications not allowed in this study,
10. previously participated in and/or were terminated from the study,
11. have a diagnosis of bipolar disorder, schizophrenia, other psychotic disorder or alcohol/substance use disorder, and/or
12. have a medical condition or are taking medications that are contraindicated for sertraline

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Treatment Engagement | 6 weeks
Treatment Adherence | 18 weeks

SECONDARY OUTCOMES:
Treatment Response | 12 weeks
Treatment Remission | 12 weeks
Maternal functional assessment | 12 weeks
Maternal healthcare utilization | 18 weeks
Infant healthcare utilization | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Linda H Chaudron, MD, MS, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States